CLINICAL TRIAL: NCT00522535
Title: Prospective Aneurysm Trial: High Angle Aorfix™ Bifurcated Stent Graft
Acronym: PYTHAGORAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lombard Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PYTHAGORAS
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: AAA; Abdominal Aortic Aneurysms; Endovascular; EVAR; Aorta; Stent Graft; Stent; Tortuous; High Angle; Angled Necks
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Open Surgical Repair (Active Comparator): Open surgical repair of abdominal aortic aneurysm. All patient enrollment and 2-year follow-ups completed.
  Interventions: Procedure: Open surgical repair
- Endovascular Repair (Experimental): Endovascular treatment arm of 160 patients having suitable anatomy for the Aorfix™ AAA Flexible Stent Graft System. Use of stent grafts in aortic angles greater than 60° has not been approved for other devices available in the US. As a result, a minimum of 120 patients in this arm will have an aortic angle between 60° and 90°.
  Patient recruitment completed; 5-year follow-up evaluations continue.
  Interventions: Device: Stent Graft
- Continued Access (Experimental): Endovascular treatment arm of 50 patients maximum having suitable anatomy for the Aorfix™ AAA Flexible Stent Graft System. This Arm will provide active sites with ongoing device access while FDA reviews the PMA.
  Patient recruitment completed; 5-year patient follow-ups continue.
  Interventions: Device: Stent Graft

INTERVENTIONS:
Procedure: Open surgical repair — Open surgical repair of abdominal aortic aneurysm
  Arms: Open Surgical Repair
Device: Stent Graft — Endovascular repair of abdominal aortic aneurysm (EVAR)
  Other Names: Aorfix™ stent graft; Aorfix™ AAA stent graft
  Arms: Continued Access; Endovascular Repair

SUMMARY:
Purpose of this study: The purpose of the study is to evaluate the safety and effectiveness of the Lombard Medical endovascular Aorfix™ AAA bifurcated stent graft in the treatment of abdominal aortic, aorto-iliac and common iliac aneurysms with anatomies including angled aorta, angled aneurysmal body, or both, between 0° and 90°.

Study hypothesis: The primary efficacy hypothesis is the proportion of grafts remaining free from endoleak, migration, and fracture at 12 months.

Efficacy: The 12 month, all cause mortality rate in the Aorfix™ group will be non-inferior to the 12 month, all cause mortality rate in the Open Control group.

Safety: The rates of early serious adverse events between 0 and 30 days post-operative in the Aorfix™ groups will be non-inferior to the early serious adverse event rates between 0 and 30 days post-operative in the Open Control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed abdominal aortic aneurysm > 4.5 cm in diameter, OR 4.0 cm or larger in diameter if symptomatic (i.e. pain, embolization), OR documented AAA growth of more than 5 mm within the previous 6 months, and/or including extension into common iliac artery (ies), and/or
* Iliac aneurysm greater than, or equal to 3.5 cm in maximum diameter.

Exclusion Criteria:

* Less than 21 years of age,
* Life expectancy less than 2 years,
* Pregnant,
* Religious cultural or other objection to the receipt of blood or blood products,
* Unwilling to comply with follow-up schedule,
* Unwillingness or inability to provide informed consent to both trial and procedure.
* Patients not expected to live more than 2 years from enrollment
* Patient has a ruptured aneurysm
* Aneurysm extends above renal arteries
* Proximal neck of aneurysm has significant loose thrombus associated with it
* Patient with an acute or chronic aortic dissection or mycotic aneurysm
* Patient has current non-localized infection (may be recruited following remission of the infection)
* Patient is allergic to device materials
* Patient is allergic to or intolerant of use of contrast media and cannot be exposed to suitable remedial treatment such as steroids and/or benadryl
* Patient is clinically and morbidly obese such that imaging would be severely adversely affected
* Patient has renal failure (serum creatinine > 2.5 mg/dL)
* Patient has an uncorrectable bleeding abnormality
* Patient has unstable angina
* Patient is receiving dialysis:
* Inflammatory aneurysm
* MI in last 6 months
* End stage COPD
* Patient has connective tissue disease (eg Marfan syndrome, Ehlers-Danlos syndrome)
* Significant (>80%) renal artery stenosis which cannot be readily treated

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2006-04; Primary Completion 2011-09 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Aorfix™ vs. Open Control All Cause Mortality | 1 year
  The 12 month, all cause mortality rate in the Aorfix™ group compared to all cause mortality rate in the Open Control group.

SECONDARY OUTCOMES:
Aorfix™ vs. Open Control Adverse Events | 30 days
  The rates of early serious adverse events between 0 and 30 days post-operative in the Aorfix™ groups compared to the early serious adverse event rates between 0 and 30 days post-operative in the Open Control group.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fillinger, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (38):
- United States (38):
  - UAB Vascular Surgery, Birmingham, Alabama
  - University of Arizona, Department of Surgery, Tucson, Arizona
  - Long Beach VA Healthcare System, Long Beach, California
  - UCSF Division of Vascular Surgery, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Holy Cross Hospital, Jim Moran Heart & Vascular Research Institute, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Baptist Hospital of Miami, Cardiac & Vascular Institute, Miami, Florida
  - Macon Cardiovascular Institute, Macon, Georgia
  - Methodist Heart Lung & Vascular Institute, Peoria, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - John Hopkins Bayview Medical Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Department of Vascular Surgery, Ann Arbor, Michigan
  - Michigan Vascular Group, Flint, Michigan
  - Abbott Northwestern / MHIF, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Dartmouth - Hitchcock Medical, Lebanon, New Hampshire
  - Englewood Hospital & Medical Center, Englewood, New Jersey
  - Newark-Beth Israel Medical Center, Newark, New Jersey
  - Albany Medical Center, Albany, New York
  - New York Presbyterian-Columbia University Medical Center Division of Vascular Surgery, New York, New York
  - Jobst Vascular Center, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pinnacle Health Hospitals, Harrisburg, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Moffitt Heart and Vascular Group, Wormleysburg, Pennsylvania
  - Sanford Clinic Clinical Research, Sioux Falls, South Dakota
  - University of Tennessee, Chattanooga, Tennessee
  - DeBakey Heart Center, Methodist Hospital, Houston, Texas
  - Sentara Heart Hospital - Vascular & Transplant Specialists, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - University of Wisconsin School of Medicine & Public Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang S, Hicks CW, Malas MB. Neck diameter and inner curve seal zone predict endograft-related complications in highly angulated necks after endovascular aneurysm repair using the Aorfix endograft. J Vasc Surg. 2018 Mar;67(3):760-769. doi: 10.1016/j.jvs.2017.07.114. Epub 2017 Sep 21. PMID 28943010
- [Derived] Malas MB, Hicks CW, Jordan WD Jr, Hodgson KJ, Mills JL Sr, Makaroun MS, Belkin M, Fillinger MF; PYTHAGORAS Investigators. Five-year outcomes of the PYTHAGORAS U.S. clinical trial of the Aorfix endograft for endovascular aneurysm repair in patients with highly angulated aortic necks. J Vasc Surg. 2017 Jun;65(6):1598-1607. doi: 10.1016/j.jvs.2016.10.120. Epub 2017 Feb 9. PMID 28190716
- [Derived] Malas MB, Jordan WD, Cooper MA, Qazi U, Beck AW, Belkin M, Robinson W, Fillinger M. Performance of the Aorfix endograft in severely angulated proximal necks in the PYTHAGORAS United States clinical trial. J Vasc Surg. 2015 Nov;62(5):1108-17. doi: 10.1016/j.jvs.2015.05.042. Epub 2015 Aug 28. PMID 26321596
- See also: Lombard Medical Technologies Inc. Homepage — http://www.lombardmedical.com